CLINICAL TRIAL: NCT03972891
Title: Influence of a Intervention Break on a Treated Phonological Process in Spontaneous Speech Situations in Children Aged 5 to 6 Years With Phonologically Delayed Development
Brief Title: Influence - Intervention Break - Children - Speech Sound Disorders
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the changed working conditions in the participating institutions after the covid-19- pandemic, the clientele of the institutions has changed. Therefore, the calculated number of cases cannot be achieved in the planned study.
Sponsor: University of Applied Sciences for Health Professions Upper Austria (Other)
Collaborators: Caritas Austria (Unknown); Volkshilfe Upper Austria (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A-2019-035
Record Dates: First submitted 2019-05-13; First posted 2019-06-04 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Speech Sound Disorder
Keywords: speech sound disorders; children
MeSH Terms: conditions — Speech Sound Disorder

STUDY DESIGN:
Intervention Model Description: Study Design: randomized control trial, single-blinded Time Perspective: prospective
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: An independent biometrician created forty envelopes (i.e., 20 blue and 20 white envelopes) for group allocation. Each envelope was filled with the group assignment ("intervention break" or "continuous therapy") and signed by the biometrician. White envelopes will only be used when all blue envelopes are opened to ensure that 20 group-balanced children can be used for interims analysis. Each envelope pack (white & blue) consisted of 10 intervention ("therapy break") and control ("continuous therapy") groups. The group allocation take place after inclusion of the child in the study. The non-transparent envelope is randomly drawn and opened by the speech therapist. The randomisation result, the name of the child and the date of the assignment will be documented in the case report form (CRF). The CRFs and the envelop will be handed over to the study director at regular intervals, whereby the biometrician is not informed about the allocation of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12-weeks intervention break (Experimental): The intervention break starts as soon as 70 - 80 % of the target phoneme / target consonant cluster can be pronounced correctly in spontaneous speech situations during therapy. The intervention break will last for 12 weeks.
  Interventions: Other: intervention break of 12 weeks
- traditional therapy (No Intervention): After 70 - 80 % of the target phoneme / target consonant cluster can be pronounced correctly in spontaneous speech situations during therapy, the children will maintain their traditional therapy until more than 90% of the target phoneme / target consonant cluster can be pronounced correctly in spontaneous speech situations (max. 12 weeks).

INTERVENTIONS:
Other: intervention break of 12 weeks — The intervention of this study is a break of the intervention for 12 weeks under the following conditions:
  * no therapeutic intervention during the break
  * no language-specific specific exercises
  * language-specific strategies in everyday life can be applied, e.g. modeling techniques
  Arms: 12-weeks intervention break

SUMMARY:
Many of the children with speech and language disorders have speech sound disorders. In German-speaking countries, it is estimated that around 16% of children between the ages of three and eight are affected by school entry. The treatment of speech sound disorders aims to enable the transfer of the learned into spontaneous speech. The purpose of this study is to ascertain, whether children, by means of a break in therapy, succeed in transferring, the target phoneme or target consonant cluster - from a certain threshold - to spontaneous language. The researchers compare the effect of the transfer to spontaneous speech situations by means of a twelve-week break from therapy with a continuous therapy.

In addition, the researchers would like to find out whether the acquisition of the grapheme has an additional positive influence on the generalization of the target phoneme or target consonant cluster in spontaneous speech situations.

The researchers also seek to understand individual differences in the generalization effects on the production of the target phoneme / target consonant cluster in spontaneous speech situations, in which the researchers document and evaluate information on the treatment method and treatment duration before the therapy break.

DETAILED DESCRIPTION:
Early detection of language development disorders and a timely delivery of appropriate measures derived from it, can prevent secondary consequences of language learning disorders. In particular, phonologically delayed disorders can have an impact on the development of literacy and place the child at risk of dyslexia. With this knowledge, that early detection and the appropriate measures derived from it can prevent the secondary consequences of a speech sound disorder, speech and language therapists strive to carry out an effective therapeutic process based on the International Classification of Functioning, Disability and Health (ICF). In the field of effectiveness research, there is consensus that the objective, which is tailored to the disorder, is closely linked to the chosen therapeutic method. Therapeutic ICF-oriented measures should be adapted to the needs of the child. Based on the current knowledge, no therapy concept can offer this, if it is used exclusively.

In effectiveness research, disagreement prevails in the area of treatment intensity and the intervention period. The therapy intensity is determined by three factors: number of properly implemented teaching episodes per session (dose), task or activity within which the teaching episodes are delivered (dose form) and the number of sessions per unit of time (e.g. once a week/once a month), It should be noted that the threshold at which speech therapy is still effective and where the intervention period is too short has mostly been derived from observations. It seems that a certain amount of developmental time is required for the consolidation of new skills. It has so far only been stated that the duration of intervention cannot be generalized for each child and that an improvement in the functional capacity of the linguistic output may be between 12 and 20 hours of intervention. In addition to the uncertainty of how high the intensity of therapy must be in order to achieve generalization effects, there is no information in science to date as to which baseline level has to be achieved for it.

Therefore the desire for systematic studies on the question: Which baseline level does a child have to reach in order to transfer the treated phonological process to the spontaneous speech during the therapy break? prevails.

Aim 1 will determine whether a 12-week intervention break in children between the ages of five and six with phonologically delayed development of one phonological process will lead to significant improvements in the transfer of the target phoneme / target consonant cluster in spontaneous speech. On the condition that the threshold of 70-80% correct pronunciation of the target phoneme / target consonant cluster was attained.

Aim 2 will determine whether children, who at the end of the therapy, do not demonstrate 100 percent correct pronunciation of the targeted phoneme / the target consonant cluster in spontaneous speech by acquiring the grapheme/graphemes (the affected treated phoneme / the affected treated consonant cluster) see an improvement of the target phoneme / target consonant cluster in spontaneous speech?

ELIGIBILITY:
Inclusion Criteria:

Speech therapists:

* Written consent to participate in the study after prior written and oral education
* At least 2 years activity in the field of children's speech therapy / therapy of infantile speech sound disorders with sufficient practical experience

Children:

* Phonological delay of one of these phonological process: palatal fronting / sch / to / s / or / ch / to / s /, velar fronting / k g / to / t d / or contact assimilation / dr / to / gr kr / and max. two phonological processes
* The treated sound can be formed correctly during therapy in the spontaneous speech situations to 70 - 80%
* The phonological process has not yet been treated by another colleague (the therapy should be carried out by a speech therapist from the beginning)
* Parental participation is given (recorded in the regular therapeutic process via anamnesis interview)
* Therapy frequency: regular once a week, but at least once every 2 weeks (so that short-term outages due to illness do not lead to exclusion from the study)
* Physiologically developed prescriptive skills
* almost native German language skills
* Written consent of the parent or guardian to participate in the study after previous oral and written information

Exclusion Criteria:

Speech therapists:

* Lack of written consent
* Practical experience in the field of children's speech therapy / therapy of infantile speech sound disorders of less than 2 years

Children:

* Younger than 5 years of age
* Therapy sounds are less than 70% correct in a spontaneous speech situation
* Inconsistent phonological disorder
* Consistent phonological disorder
* Childhood apraxia of speech
* Myofunctional disorders
* Isolated articulation disorder (e.g. lateral or interdental articulation)
* Auditory processing disorders
* Disorders of speech understanding
* Autism spectrum disorders
* Cognitive developmental disorders
* Deficits in prescriptive skills
* Missing written consent of the parents

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Changes in the target phoneme / target consonant cluster accuracy in spontaneous speech situations within-group | 12-week
  The phoneme accuracy will be determined by a standardised diagnostic assessment for speech sound disorders, a single-word test (PLAKKS), and by elicited a continuous speech sample (non-standardized assessment) für 15 minutes. For the speech sample the researchers will use the same situation pictures in a play situation for all test times to allow for direct comparison.
Changes in the target phoneme / target consonant cluster accuracy in spontaneous speech situations within-group/in group interaction | 12-week
  The phoneme accuracy will be determined by a standardised diagnostic assessment for speech sound disorders, a single-word test (PLAKKS), and by elicited a continuous speech sample (non-standardized assessment) für 15 minutes. For the speech sample the researchers will use the same situation pictures in a play situation for all test times to allow for direct comparison.

SECONDARY OUTCOMES:
Changes in the target phoneme/ consonant cluster accuracy in spontaneous speech situations within-group | 1 - 2 weeks after the target grapheme has been learned in school (0.5 - 3.5 months after school entry)
  The phoneme accuracy will be determined by a standardised diagnostic assessment for speech sound disorders, a single-word test (PLAKKS), and by elicited a continuous speech sample (non-standardized assessment) für 15 minutes. For the speech sample the researchers will use the same situation pictures in a play situation for all test times to allow for direct comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Detter-Biesl, MSc, Study Director — University of Applied Sciences for Health Professions Upper Austria
Locations (1):
- Caritas Österreich, Caritas für Kinder und Jugendliche, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoder P, Fey ME, Warren SF. Studying the impact of intensity is important but complicated. Int J Speech Lang Pathol. 2012 Oct;14(5):410-3. doi: 10.3109/17549507.2012.685890. Epub 2012 May 31. PMID 22646316
- [Background] Warren SF, Fey ME, Yoder PJ. Differential treatment intensity research: a missing link to creating optimally effective communication interventions. Ment Retard Dev Disabil Res Rev. 2007;13(1):70-7. doi: 10.1002/mrdd.20139. PMID 17326112
- [Background] Baker E. Optimal intervention intensity in speech-language pathology: discoveries, challenges, and unchartered territories. Int J Speech Lang Pathol. 2012 Oct;14(5):478-85. doi: 10.3109/17549507.2012.717967. PMID 22974107
- [Background] Allen MM. Intervention efficacy and intensity for children with speech sound disorder. J Speech Lang Hear Res. 2013 Jun;56(3):865-77. doi: 10.1044/1092-4388(2012/11-0076). Epub 2012 Dec 28. PMID 23275415
- [Background] Williams AL. Intensity in phonological intervention: is there a prescribed amount? Int J Speech Lang Pathol. 2012 Oct;14(5):456-61. doi: 10.3109/17549507.2012.688866. Epub 2012 Jun 11. PMID 22686582